CLINICAL TRIAL: NCT03918798
Title: Randomized, Multi-center, Double-blind, Two-armed, Parallel Active Groups, Prospective Trial, to Evaluate, in Pediatric Population, the Efficacy and Safety of Chloroprocaine 1% and 2% for Peripheral Nerve Block.
Brief Title: The Efficacy and Safety of Chloroprocaine 1% and 2% in Pediatric Population
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sintetica SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CHL.2/04-2015
Record Dates: First submitted 2019-03-20; First posted 2019-04-18 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Hernia, Inguinal; Flat Foot
Keywords: Surgery; Hernia, Inguinal; Flat Foot; Pediatric population; Peripheral nerve block
MeSH Terms: conditions — Hernia, Inguinal; Flatfoot | interventions — chloroprocaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chloroprocaine 1% (Experimental): All the eligible patients will be administrated by Chloroprocaine 1 % according to the randomization criteria.
  Interventions: Drug: Chloroprocaine 1% Injectable Solution
- Chloroprocaine 2% (Experimental): All the eligible patients will be administrated by Chloroprocaine 2 % according to the randomization criteria.
  Interventions: Drug: Chloroprocaine 2% Injectable Solution

INTERVENTIONS:
Drug: Chloroprocaine 1% Injectable Solution — All the eligible patients will be administrated by Chloroprocaine 1 % according to the randomization criteria.
  Other Names: ARM 1
  Arms: Chloroprocaine 1%
Drug: Chloroprocaine 2% Injectable Solution — All the eligible patients will be administrated by Chloroprocaine 1 % according to the randomization criteria.
  Other Names: ARM 2
  Arms: Chloroprocaine 2%

SUMMARY:
Randomized, multi-center, double-blind, two-armed, parallel active groups, prospective trial to evaluate the efficacy and safety of local anesthetic Chloroprocaine at two different concentrations ( at 1% and 2%) in a pediatric population subjected to peripheral nerve block due to Inguinal hernia repair or Flat foot surgery. The present Protocol is part of an extensive Pediatric Investigational Plan (PIP) in the contest of the marketing authorization application of chloroprocaine use for perineural block. The PDCO has adopted a positive opinion.

DETAILED DESCRIPTION:
Randomized, multi-center, double-blind, two-armed, parallel active groups, prospective trial, to evaluate, in pediatric population undergoing Flat Foot surgery or Inguinal hernia repair, the efficacy and safety of chloroprocaine 1% and 2% for peripheral nerve block (PNB) based on concentration-response relationships. The present protocol is part of an extensive Pediatric Investigational Plan (PIP) which has been submitted to the Paediatric Committee (PDCO) of the European Medicine Agency (EMA)in the contest of the marketing authorization application of chloroprocaine use for perineural block. The PDCO has adopted a positive opinion on both the PIP and the present clinical protocol.

Chloroprocaine Hydrochloride 1% Sintetica is currently marketed in 9 European countries as intrathecal (spinal) anesthetic in adults where the planned surgical procedure is not expected to exceed 40 minutes. Since 2015, the Marketing Authorization in Switzerland has been extended to chloroprocaine HCl 20 mg/mL and 30 mg/mL solutions for injection, for local anesthesia by infiltration, for PNB and epidural block, respectively. Regional analgesia, and specifically PNB, is an acceptable means of providing intraoperative anesthesia and postoperative analgesia in neonates, infants, and children while decreasing the use of systemic opioids and avoiding opioid-related adverse effects. With the advent of ultrasound and improvements in equipment in the last decade, the utilization of PNB in children has increased tremendously.

Flat Foot and inguinal hernia repair have been considered the ideal surgeries for testing the clinical efficacy and safety of chloroprocaine since they are short procedures with low postoperative pain that only require a short- to intermediate-acting agent. The study consists of a treatment period of 1 day and of a single perineural injection, administered through ultrasound-guided technique in order to avoid the risk of chloroprocaine IV injection. A total of 174 (87 per treatment group, allocated to 1% or 2% arm in a ratio of 1:1) male and female paediatric patients (age range from birth to <18 years) undergoing Flat Foot surgery or Inguinal hernia repair, planned for peripheral nerve block anaesthesia and equally distributed within the two surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female paediatric patients from birth to <18 years scheduled for:

   * Flat Foot surgery (6 to <18 years; children and adolescents)planned for sciatic nerve block short-lasting anaesthesia,
   * inguinal hernia repair (28 day from birth to 6 years; infants-toddlers and children)planned for ilioinguinal/iliohypogastric block short-lasting anaesthesia;
2. Normally active and otherwise judged to be in good health on the basis of medical history, physical examination, with normal lean body mass (BMI18,5 - 24,9 Kg/m2 inclusive) and normal body development (normal weight and height according to local paediatric Height and Weight Chart);
3. ASA I and ASA II patients;
4. Written informed consent provided by parents/tutor, willing and able to understand the purpose of the study, including possible risks and side effects, and willing and able to comply, on their behalf and of the minor, with the study requirements;
5. Willing and able to give additional written informed consent by itself, in case of children and adolescents, in addition to parents/tutor;
6. Willing and able, in case of children and adolescents, to comply with the study requirements on their behalf.

Exclusion Criteria:

1. ASA > II patients;
2. Preexistent infection at injection site;
3. Use of opioids, antidepressants, anticonvulsant, sulfonamide, vasopressors, ergot-type oxytocic drug and mixtures of local anaesthetics, antiarrhythmic drug class III, such as amiodarone, strong inhibitors of CYP1A2, such as fluvoxamine and enoxacin;
4. Use of medication(s) known to interfere with the extent of regional blocks for 2 weeks before the start of the study;
5. History of drug or alcohol abuse;
6. Sensitivity among the study medication active ingredient, the members of the PABA esters group and amides-type local anesthetic group;
7. Clinical history of allergy, hypersensitivity or intolerance to the study medication or other medications used during surgery;
8. Pregnancy and lactation: positive pregnancy test at screening (if applicable), pregnant or lactating (the pregnancy test will be performed to all fertile subset);
9. Participation in any other clinical study within the 3 months prior to the screening.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 174 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall proportion of patients, in each of the two dosage level groups, not requiring rescue anesthesia during surgery. | Visit 2 (Day 1; surgery/discharge)
  The primary efficacy endpoint of the study will be represented by the overall proportion of patients, in each of the two dosage level groups, not requiring rescue anesthesia during surgery.

SECONDARY OUTCOMES:
Proportion of patients, in both of the two dosage level groups, not requiring rescue anaesthesia (fentanyl) during the two surgical procedures separately | Visit 2 (Day 1; surgery/discharge); FU phone call I( 24 hrs from Visit 2); FU phone call II (7 days from Visit 2)
  Proportion of patients, in both of the two dosage level groups, not requiring rescue anaesthesia (fentanyl) during the two surgical procedures separately; Time to onset of sensory block, defined as the time period from completion of the injection (time 0 min) to the achievement of complete sensory block, assessed by pinprick test associated with heart rate measurement, and evaluated for both surgeries; Time to regression of motor block evaluated in 'calcaneo stop' surgery only and assessed by a grade I of the standard Bromage scale (i.e. free movement of legs and feet). Pain intensity evaluated five times in the first 3 hours after patient's awakening andduring the home discharge visit (V2). The technique and appropriate scale for pain measurement are age-dependent therefore, different tools will have to be used for the evaluation: COMFORT scale for patients <2 months of age; FLACC scale for patients aged _ 2 months _ 6 years; Wong-Baker scale for patients over 6 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Mosetti, MD, Principal Investigator — Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Locations (9):
- Italy (7):
  - Ospedale Pediatrico Bambin Gesù di Roma Dipartimento di Emergenza Accettazione (DEA) e A.R.C.O, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli U.O.C. Anestesia delle Chirurgie Generali del Policlinico, Rome, Lazio
  - Ospedale San Raffaele Anestesia e Rianimazione del distretto testacollo, Milan, Lombardy
  - Ospedale Infantile Santa Margherita di Torino Anestesia e Rianimazione Pediatrica, Turin, Piedmont
  - Ospedale Universitario Santa Maria della Misericordia S.C. di Anestesia e Rianimazione 2, Perugia, Umbria
  - Ospedale Pediatrico Giovanni XXIII, Bari
  - ASST Gaetano Pini CTO, Milan
- Spain (2):
  - Consorcio Hospital General Universitario De Valencia Cirugía Mayor Ambulatoria Y Cirugía General Y Del Aparato Digestivo, Valencia
  - Hospital Universitario Y Politecnico La Fe Cirugía Pediátrica Avda. Fernando Abril, Valencia

IPD SHARING:
Plan to Share IPD: No
It is not yet known if there will be a plan to make IPD available.

DOCUMENTS (3):
  • Study Protocol (2018-06-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT03918798/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-25): https://cdn.clinicaltrials.gov/large-docs/98/NCT03918798/SAP_002.pdf
  • Informed Consent Form (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/98/NCT03918798/ICF_001.pdf